CLINICAL TRIAL: NCT01135862
Title: Platelet Administration To Patients With Traumatic Brain Injury Who Were Treated With Aspirin
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Tel-Aviv Sourasky Medical Center (Other Government)
Responsible Party: Department of Neurosurgery, Tel Aviv Sourasky Medical Center
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CTIL-000-JR-08-TASMC
Record Dates: First submitted 2010-03-08; First posted 2010-06-03 (Estimated); Last update posted 2010-06-03 (Estimated); Status verified 2010-06

CONDITIONS: Aspirin Treatment; Traumatic Intracranial Bleed; Hemorrhage Growth; Neurological Outcome
MeSH Terms: interventions — Platelet Count

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- platelet administered (Experimental): patients will receive 6 packs of platelets
  Interventions: Drug: platelets
- no platelets administered (No Intervention): patients will not receive platelets
  Interventions: Drug: platelets

INTERVENTIONS:
Drug: platelets — 6 packs of platelets will be administered

SUMMARY:
Traumatic brain injury (TBI) is a devastating disease with high morbidity and mortality. Although not fully proved, it is commonly accepted that the morbidity and mortality and proportional to the extent of intracranial bleeds (i.e. - larger hemorrhages cause more injury than smaller ones).

Aspirin is a commonly used antiaggregate drug that interferes with the clotting system. The antiaggregate effect may be neutralized by administration of platelets. Thus, potentially, patients receiving Aspirin and undergoing TBI, are at a higher risk for increasing an intracranial bleed.

In this prospective study, the investigators randomize patients receiving aspirin that have a traumatic intracranial bleed to two groups, one - that will receive platelets, and the other that will not receive platelets.

The primary end point of the study is to evaluate the effect of platelet administration of the enlargement of traumatic intracranial bleeds, and try and evaluate any clinical outcome differences between the two groups.

DETAILED DESCRIPTION:
Traumatic brain injury (TBI) is a devastating disease with high morbidity and mortality. Although not fully proved, it is commonly accepted that the morbidity and mortality and proportional to the extent of intracranial bleeds (i.e. - larger hemorrhages cause more injury than smaller ones).

Aspirin is a commonly used antiaggregate drug that interferes with the clotting system. The antiaggregate effect may be neutralized by administration of platelets. Thus, potentially, patients receiving Aspirin and undergoing TBI, are at a higher risk for increasing an intracranial bleed.

In this prospective study, we randomize patients receiving aspirin that have a traumatic intracranial bleed to two groups, one - that will receive platelets, and the other that will not receive platelets.

The primary end point of the study is to evaluate the effect of platelet administration of the enlargement of traumatic intracranial bleeds, and try and evaluate any clinical outcome differences between the two groups.

ELIGIBILITY:
Inclusion Criteria:

* age >18 years old
* chronic aspirin treatment
* first CT scan less than 12 hours following the trauma
* GCS >3
* no immediate surgical cranial lesion
* isolated head injury
* consent
* contusions >1.5cc or acute subdural hemorrhage in any size

Exclusion Criteria:

* anticoagulation treatment
* more than one antiaggregate
* coagulopathy
* thrombocytopenia (less than 100000)
* intracranial tumor
* active hematological disease
* more than 8 hours between first and second CT scan
* more than 2 hours between first CT and platelet admission

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2010-06; Primary Completion 2011-06 (Estimated); Study Completion 2013-06 (Estimated)

PRIMARY OUTCOMES:
efficacy of platelet administration in lowering the rate of early hemorrhagic growth within 6 hours | 6 hours
are lower aspirin doses a risk for early hemorrhagic growth | 6 hours

SECONDARY OUTCOMES:
vascular complications | within 1 month from platelet admission
  vascular complications include active ischemic heart disease (MI, unstable angina), ischemic stroke, acute peripheral vasculopathy, deep vein thrombosis, and pulmonary emboli these complications will be diagnosed clinically and not by screening procedures.
complications attributed to platelets as listed below | within 1 week
  these complications include an exacerbation of congestive heart failure, or any allergic reaction to platelet admission such as fever, rigor, rash, hemodynamic collapse occuring within 6 hours of platelet admission.
  other events which will be attributed to platelet admission are sepsis <48 hours after platelet admission or new thrombocytopenia occurring within 1 week after admission of platelets.
difference in neurological outcome between both groups | 1 month, 6 months, and 1 year after the traumatic brain injury
  as evaluated by Glasgow Outcome Score (GOS)

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan Roth, MD, Principal Investigator — Tel-Aviv Sorasky Medical Center
Locations (1):
- Tel-Aviv Sourasky Medical Center, Tel Aviv, Israel